CLINICAL TRIAL: NCT04803591
Title: Efficacy of Tranexamic Acid in Femoral Shaft Fractures Osteosynthesis; A Double Blind Randomized Controlled Trial
Brief Title: This is a Study to Verify if Tranexamic Acid Can Reduce the Anemia After a Femoral Shaft Fractures Surgery
Acronym: ORL-ORT-023
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not approved by Ethics Commettee
Sponsor: Christian Candrian (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL - ORT - 023
Record Dates: First submitted 2021-03-10; First posted 2021-03-17 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Femoral Shaft Fracture
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: Tranexamic Acid group (Experimental): Patients in the Tranexamic Acid (TXA) group (arm-A) will be administered with 2 doses of intravenous tranexamic acid (cumulative dose 10ml=1g) as follows: the first dose 10 minutes before the surgical incision (1 vial of 5 ml = 0,5g by slow intravenous injection(=1ml/minute)), and the second 3 hours after the start of surgery (1 vial of 5 ml = 0,5g, by slow intravenous injection).
  Interventions: Drug: Tranexamic Acid
- B : No treatment group (No Intervention): In the control group, will not be administered TXA or any other drugs.

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic Acid will be administered as an injectable solution (500mg/5ml or 1000mg/10ml).
  Other Names: TRANEXAM OrPha Inj Lös 500 mg/5ml
  Arms: A: Tranexamic Acid group

SUMMARY:
The investigators are going to evaluate if adding Tranexamic Acid in femoral shaft fractures surgery can lead to any advantages to the participants, namely if it can reduce post-operative anaemia, blood loss, blood transfusion requirements, length and cost of hospitalisation.

DETAILED DESCRIPTION:
Lower limb procedures represent the majority of orthopaedic surgeries, including joint arthroplasties, sport medicine treatments, and fractures osteo-synthesis, with a rate over 500 per 100,000 population every year, increasing. Albeit being successful procedures routinely performed in the clinical practice, they are frequently encumbered by complications. In particular, femur fractures are common and frequently result in considerable blood loss, ranging from 900 to 1,500 ml, which exposes patients to postoperative anaemia and reduced functional recovery. Allogenic blood transfusions are financial burden, and, even more, they are associated with an unneglectable risk of serious complications, including infection, immuno-suppression, cardiovascular dysfunction, resulting in potentially life-threatening effects on patients. Various strategies have been attempted to minimize blood loss and the need for blood transfusion, and to this aim the use of hemostatic agents, in particular of tranexamic acid (TXA), has recently widely increased in orthopaedic lower limb surgery.

TXA is a synthetic anti-fibrinolytic agent that competitively blocks the lysine binding sites on plasminogen, thereby slowing the conversion of plasminogen to plasmin, thus preventing fibrin clot degradation. A large amount of randomized controlled trials and meta-analysis converge in showing that TXA, applied either through systemic or local administration, is effective in reducing blood loss and subsequent transfusions in lower limb fractures surgery, especially in hip fracture patients, as well in replacement procedures. However, there are still concerns about the risk of increasing venous thromboembolic (VTE) complications, such as deep venous thrombosis or pulmonary embolisms; overall, the scientific high-level literature evidence supports the safety of TXA for the different orthopaedic applications.

This is a 2-arm study aimed at comparing the Tranexamic Acid supplementation protocol and evaluating his advantages over routine protocols. The primary objective will be the effect on postoperative anaemia, detected by serial measurements of haemoglobin, of TXA supplementation for femoral shaft fractures surgery. The secondary objectives of the study will be the comparison between I.V. peri-operative TXA supplementation and normal protocol without TXA in terms of post-operative anaemia (detected by serial haematocrit measurements), intra-operative blood loss, post-operative blood loss, total blood loss (evaluated using the Hb balance formula, estimated blood loss, blood transfusion requirements, length of hospitalisation, cost-effectiveness and frequency of adverse events. In particular the study aims to assess safety of TXA and its tolerability in terms of incidence of venous thromboembolic complications, such as deep venous thrombosis or pulmonary embolisms, wound infection, and death. The safety of TXA supplementation protocol will be verified comparing to the no-treatment group in terms of incidence of complications, such as deep venous thrombosis (based on the Homan sign and Mose sign and confirmed by compression ultrasonography upon clinical suspicion), Pulmonary embolism (confirmed by spiral computed tomography), cerebrovascular accident (confirmed by computed tomographic scan or magnetic resonance imaging), and acute coronary syndrome or myocardial infarction (confirmed by troponin I estimation and electrocardiogram changes), infection, and death. This randomized control trial will thus define if the peri-operative protocol should be implemented with tranexamic acid to reduce post-operative anaemia and blood loss and the rate of blood transfusion leading to a better cost effectiveness, without an increase in adverse events.

The study presents only minimal risks for the included patients.

ELIGIBILITY:
Inclusion Criteria:

* Acute femoral shaft fracture.
* Patients treated surgically with intramedullary nail or femoral plate
* Patients aged 18-80 years old.
* Patients with a BMI >18.5 and <35.
* Patients able to provide informed consent and follow all the study procedures as indicated by the protocol.
* Informed Consent as documented by signature

Exclusion Criteria:

* Pathological fracture or other lower limb fractures associated or multiple fractures.
* Use of any anticoagulant at the time of admission (eg, vitamin K antagonists, anti-thrombin agents, antiplatelet agents or factor IIa and Xa inhibitors).
* Contraindications to TXA (eg documented allergy to TXA).
* Hepatic dysfunction (aspartate transaminase (AST)/alanine transaminase (ALT)>60 U/l) or renal dysfunction (Cr >1.5 mg/dl of glomerular filtration rate (GFR)>30 ml/min).
* History of DVT or pulmonary embolus.
* Active coronary artery disease or cerebrovascular accident (event in the past 12 months).
* Coagulopathy based on admission laboratory values (international normalised ratio (INR)>1.4, partial thromboplastin time (PTT)>1.4× normal sec, platelets <50 000 per mm3)
* Women who are pregnant or breast feeding.
* Known or suspected non-compliance, drug or alcohol abuse.
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant.
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative anaemia | 3 days after surgery
  Postoperative anaemia detected by daily measurements of haemoglobin in the first 3 days after surgery

SECONDARY OUTCOMES:
Post-operative anaemia | 3 days
  Post-operative anaemia reported as changes in haemoglobin and haematocrit values during the first 3 days after surgery.
Intra-operative blood loss | Day 0
  This outcome will be documented using a suction apparatus during the procedure. Blood collected in the suction bottle will be measured by subtracting the volume of saline used for wash.
Post-operative blood loss at during the first 2 days after surgery | Up to day 2
  This outcome will be documented using postoperative drain outputs. Blood collected in the drain outputs will be measured in milliliter at 24h and 48h
Estimated total blood loss. | Up to day 2
  This outcome will be documented using Hb balance formula.
Estimated total blood loss. | Up to day 2
  This outcome will be documented using Gross Formula.
Blood transfusion requirements. | Up to day 2
  This outcome will be documented in terms of number of patients who required packed red blood cell (PRBC) (transfusion rate) and the mean number of transfusion units per patient during all the length of hospitalization.
Length of hospital stay | Up to week 2
  Length of hospital stay
Cost effectiveness of the treatment with tranexamic acid. | 1 week
  This outcome will be documented reporting the mean cost per patient as sum of the cost TXA administration (if administered), the transfusion cost per patients, and the cost of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, MD; Prof., Principal Investigator — EOC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Haghighi M, Ettehad H, Mardani-Kivi M, Mirbolook A, Nabi BN, Moghaddam R, Sedighinejad A, Khanjanian G. Does Tranexamic Acid Reduce Bleeding during Femoral Fracture Operation? Arch Bone Jt Surg. 2017 Mar;5(2):103-108. PMID 28497100
- [Background] Gross JB. Estimating allowable blood loss: corrected for dilution. Anesthesiology. 1983 Mar;58(3):277-80. doi: 10.1097/00000542-198303000-00016. No abstract available. PMID 6829965
- [Background] Drakos A, Raoulis V, Karatzios K, Doxariotis N, Kontogeorgakos V, Malizos K, Varitimidis SE. Efficacy of Local Administration of Tranexamic Acid for Blood Salvage in Patients Undergoing Intertrochanteric Fracture Surgery. J Orthop Trauma. 2016 Aug;30(8):409-14. doi: 10.1097/BOT.0000000000000577. PMID 26978136
- [Background] Nagra NS, van Popta D, Whiteside S, Holt EM. An analysis of postoperative hemoglobin levels in patients with a fractured neck of femur. Acta Orthop Traumatol Turc. 2016 Oct;50(5):507-513. doi: 10.1016/j.aott.2015.11.001. Epub 2016 Oct 15. PMID 27756504
- [Background] Lua J, Tan VH, Sivasubramanian H, Kwek E. Complications of Open Tibial Fracture Management: Risk Factors and Treatment. Malays Orthop J. 2017 Mar;11(1):18-22. doi: 10.5704/MOJ.1703.006. PMID 28435569
- [Background] Neumann MV, Strohm PC, Reising K, Zwingmann J, Hammer TO, Suedkamp NP. Complications after surgical management of distal lower leg fractures. Scand J Trauma Resusc Emerg Med. 2016 Dec 9;24(1):146. doi: 10.1186/s13049-016-0333-1. PMID 27938394
- [Background] Maniar RN, Kumar G, Singhi T, Nayak RM, Maniar PR. Most effective regimen of tranexamic acid in knee arthroplasty: a prospective randomized controlled study in 240 patients. Clin Orthop Relat Res. 2012 Sep;470(9):2605-12. doi: 10.1007/s11999-012-2310-y. Epub 2012 Mar 15. PMID 22419350
- [Background] Jiang W, Shang L. Tranexamic acid can reduce blood loss in patients undergoing intertrochanteric fracture surgery: A meta-analysis. Medicine (Baltimore). 2019 Mar;98(11):e14564. doi: 10.1097/MD.0000000000014564. PMID 30882622
- [Background] Xin WQ, Gao YL, Shen J, Yang XY. Intravenous tranexamic acid reduces blood transfusions in revision total hip arthroplasty: a meta-analysis. J Comp Eff Res. 2019 Aug;8(11):917-928. doi: 10.2217/cer-2019-0030. Epub 2019 Aug 22. PMID 31436114
- [Background] Yao RZ, Gao WQ, Wang BW, Wang GL, Wu CX, A-Mu YD. Efficacy and Safety of Tranexamic Acid in Reducing Blood Loss of Lower Extremity Osteotomy in Peri-acetabulum and High Tibia: A Systematic Review and Meta-analysis. Orthop Surg. 2019 Aug;11(4):545-551. doi: 10.1111/os.12515. PMID 31456323
- [Background] Chen S, Wu K, Kong G, Feng W, Deng Z, Wang H. The efficacy of topical tranexamic acid in total hip arthroplasty: a meta-analysis. BMC Musculoskelet Disord. 2016 Feb 16;17:81. doi: 10.1186/s12891-016-0923-0. PMID 26878845
- [Background] Moskal JT, Capps SG. Meta-analysis of Intravenous Tranexamic Acid in Primary Total Hip Arthroplasty. Orthopedics. 2016 Sep 1;39(5):e883-92. doi: 10.3928/01477447-20160526-02. Epub 2016 Jun 1. PMID 27248332
- [Background] Barrachina B, Lopez-Picado A, Remon M, Fondarella A, Iriarte I, Bastida R, Rodriguez-Gascon A, Achaerandio MA, Iturricastillo MC, Aizpuru F, Valero CA, Tobalina R, Hernanz R. Tranexamic Acid Compared with Placebo for Reducing Total Blood Loss in Hip Replacement Surgery: A Randomized Clinical Trial. Anesth Analg. 2016 Apr;122(4):986-95. doi: 10.1213/ANE.0000000000001159. PMID 26991616
- [Background] Yue C, Kang P, Yang P, Xie J, Pei F. Topical application of tranexamic acid in primary total hip arthroplasty: a randomized double-blind controlled trial. J Arthroplasty. 2014 Dec;29(12):2452-6. doi: 10.1016/j.arth.2014.03.032. Epub 2014 Mar 29. PMID 24793893
- [Background] Tengberg PT, Foss NB, Palm H, Kallemose T, Troelsen A. Tranexamic acid reduces blood loss in patients with extracapsular fractures of the hip: results of a randomised controlled trial. Bone Joint J. 2016 Jun;98-B(6):747-53. doi: 10.1302/0301-620X.98B6.36645. PMID 27235515
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146
- [Background] Good L, Peterson E, Lisander B. Tranexamic acid decreases external blood loss but not hidden blood loss in total knee replacement. Br J Anaesth. 2003 May;90(5):596-9. doi: 10.1093/bja/aeg111. PMID 12697586
- [Background] Lisander B, Ivarsson I, Jacobsson SA. Intraoperative autotransfusion is associated with modest reduction of allogeneic transfusion in prosthetic hip surgery. Acta Anaesthesiol Scand. 1998 Jul;42(6):707-12. doi: 10.1111/j.1399-6576.1998.tb05305.x. PMID 9689278
- [Background] Vaishya R, Lal H. Three common orthopaedic surgical procedures of the lower limb. J Clin Orthop Trauma. 2018 Apr-Jun;9(2):101-102. doi: 10.1016/j.jcot.2018.04.013. Epub 2018 May 4. No abstract available. PMID 29896008
- [Background] Wertheimer A, Olaussen A, Perera S, Liew S, Mitra B. Fractures of the femur and blood transfusions. Injury. 2018 Apr;49(4):846-851. doi: 10.1016/j.injury.2018.03.007. Epub 2018 Mar 7. PMID 29566986
- [Background] Lee C, Porter KM. Prehospital management of lower limb fractures. Emerg Med J. 2005 Sep;22(9):660-3. doi: 10.1136/emj.2005.024489. PMID 16113195
- [Background] Madjdpour C, Spahn DR. Allogeneic red blood cell transfusions: efficacy, risks, alternatives and indications. Br J Anaesth. 2005 Jul;95(1):33-42. doi: 10.1093/bja/aeh290. Epub 2004 Oct 14. PMID 15486006
- See also: helsinki-ethical-principles-for-medical-research-involving-human-subjects — http://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/